CLINICAL TRIAL: NCT02355730
Title: Blood Donation for the Development and Optimisation of the Second Generation Microvisk International Normalized Ratio (INR) Testing System for the Measurement of Prothrombin Time (PT)/INR in Patients on Warfarin Therapy.
Brief Title: Blood Donation From Warfarin Users for the Development of POC INR Monitor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Microvisk Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: RDE03
Record Dates: First submitted 2015-01-16; First posted 2015-02-04 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-01

CONDITIONS: Atrial Fibrillation; Pulmonary Embolism; Deep Vein Thrombosis
MeSH Terms: conditions — Atrial Fibrillation; Pulmonary Embolism; Venous Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Warfarin Patients (Experimental): Single Arm - blood collection by venepuncture in patients undergoing Warfarin Therapy
  Interventions: Procedure: Venepuncture

INTERVENTIONS:
Procedure: Venepuncture — Venepuncture to collect blood samples from Patients undergoing Warfarin Therapy.

SUMMARY:
This study is to further develop and optimise the design and manufacturing process of a handheld device to monitor and manage Warfarin (blood thinning anticoagulation drug) therapy. The device comprises of a handheld instrument and a disposable test strip and reports how blood coagulation is working in terms of standardised units called International Normalised Ratio (INR). A single drop of fresh whole blood and plasma will be added to the strip and the INR result displayed on the instrument. Blood samples are to be collected from patients attending a hospital based INR clinic who are on Warfarin Therapy. The samples are to be used in a series of experiments in the laboratory to test the Microvisk POC INR Monitors accuracy, precision, stability and robustness.

DETAILED DESCRIPTION:
The number of patients receiving anticoagulation therapy with warfarin and other vitamin K antagonists has been rising in recent years. Increasing life expectancy is increasing the proportion of the population having conditions such as Atrial Fibrillation and venous thrombosis, where primary and secondary prevention of thromboembolic complications are best achieved with anticoagulation.

Unpredictable pharmacokinetics, widespread interactions with drugs and food and the narrow therapeutic window make closely monitoring Vitamin K antagonists a necessity. Portable point of care (POC) coagulometers which measure PT from capillary whole blood and provide an INR reading within a few minutes are already widely available throughout North American and Europe. They give comparable results when compared to laboratory based systems are popular with patients and significantly shorten the duration of clinics. In addition, the United Kingdom Department of Health has been encouraging the use of anticoagulation services in Primary Care Trusts the aim being to provide INR monitoring in community clinics and General Practice surgeries relieving pressure on hospital services and reducing inconvenience for patients.

Although coagulometers are now commercially available the Microvisk INR Testing System has been designed to have advantages, particularly in terms of test robustness, user comfort, ease of use and reduction of user error. The present trial has been designed to develop the second generation Microvisk INR Test System; blood samples will also be used to optimise manufacturing processes and verify the quality of Test Strip Lots.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, greater than 18 years of age
2. Subject is receiving warfarin (or warfarin-like) therapy as part of their clinical care
3. Subject is informed and has been given ample time and opportunity to think about his/her participation and has given his/her written informed consent

Exclusion Criteria:

1. Subjects aged <18 years of age
2. Subjects who are unable to give written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1560 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The Primary Outcome will be measured in terms of differences in International Normalised Ratio when the Generation 2 system is tested against the Generation 1 system using the blood samples from the same donors. | 2 years
  The Primary Outcome will be measured in terms of differences in International Normalised Ratio when the Generation 2 system is tested against the Generation 1 system using the blood samples from the same donors. Those differences will be reported in terms of accuracy, precision and sensitivity to interferents.

SECONDARY OUTCOMES:
The Secondary Outcome will be measured in terms of differences in International Normalised Ratio when the Generation 2 system is tested against the International Standard Method using the blood samples from the same donors. | 2 years
  A master batch of test strips will be calibrated against an International Reference Preparation (rTF/09) thromboplastin. The accuracy of the master batch will be verified using patient samples.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Hock Toh, Professor, Study Chair — Royal Liverpool and Broadgreen University Hospital Trust
Locations (1):
- Royal Liverpool & Broadgreen University Hospital NHS Trust, Liverpool, Merseyside, United Kingdom